CLINICAL TRIAL: NCT03969134
Title: A Phase IIb Study to Assess the Safety, Efficacy and Immunogenicity of the Leishmania Vaccine ChAd63-KH in Post-kala Azar Dermal Leishmaniasis
Brief Title: A Study to Assess the Safety, Efficacy and Immunogenicity of Leishmania Vaccine ChAd63-KH in PKDL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of York (Other)
Responsible Party: Principal Investigator, Paul Kaye, Project Lead, University of York
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEISH2b
Record Dates: First submitted 2019-05-22; First posted 2019-05-31 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Leishmaniasis, Cutaneous
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Intervention Model Description: Randomised, double blinded, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Fifty volunteers receive a single intramuscular dose of ChAd63 KH 7.5x1010vp and 50 placebo. Investigators and the participant will be blinded. A pharmacist and nurse will prepare the injections. There will be stratification between patients aged 12-17, and patients aged 18-50, to ensure balanced randomisation. The pharmacist will be told which age strata the patient is in by a nurse, and will prepare the injection with the study nurse. There will be two series of sealed envelopes, one for each of the adolescent and adult cohorts. These envelopes will have external labelling, with the cohort, and successive cohort patient numbering. Each envelope contains randomisation to VACCINE or SALINE. The vaccine and placebo injections will be prepared in blacked-out syringes labelled with patient cohort number. The study nurse will take the prepared injection to the clinical team for administration. The syringe will be further labelled with the patient's initials, date and time of injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine arm (Active Comparator): ChAd63 KH 7.5x1010 vp, single dose, by IM injection
  Interventions: Biological: ChAd63-KH
- Placebo (Placebo Comparator): Normal Saline, single dose, by IM injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ChAd63-KH — The vaccine will be injected intramuscularly into the arm.
  Arms: Vaccine arm
Other: Placebo — The placebo will be injected intramuscularly into the arm.
  Arms: Placebo

SUMMARY:
This trial is designed to assess the therapeutic efficacy and safety of CHAd63-KH, a new candidate Leishmania vaccine, in patients with persistent PKDL. 100 participants will be randomly assigned (50 participants in each arm) to receive placebo or ChAd63-KH 7.5 x10(10)vp. Doses will be administered at a single time point.

DETAILED DESCRIPTION:
This study is a randomised, double blinded, placebo controlled trial designed to assess the therapeutic efficacy and safety of CHAd63-KH, a new candidate Leishmania vaccine, in patients with persistent PKDL. 100 participants will be randomly assigned (50 participants in each arm) to receive placebo or ChAd63-KH 7.5 x10(10)vp intramuscular injection into the deltoid region. Doses will be administered at a single time point. Volunteers aged between 12-50 years with persistent PKDL will be recruited at Professor El-Hassan's Centre for Tropical Medicine, Dooka, Gedarif State, Sudan, and will be followed up for 120 days after the dosing visit. The trial is planned to run for 24 months.

Secondary objectives are as follows:

1. To compare the humoral and cellular immune responses generated by the candidate vaccine in patients with persistent PKDL.
2. To observe any clinical changes in the cutaneous PKDL disease over a 120 day period following vaccination

ELIGIBILITY:
Inclusion Criteria:

* The volunteer must be:

  * Aged 12 to 50 years on the day of screening
  * Females must be unmarried, single, or widowed
  * Willing and able to give written informed consent
  * For adolescents aged 12 to 17 years on the day of screening written informed consent from a parent must be obtained and assent from them.

All Participants

* Uncomplicated PKDL of > 6 month's duration
* Available for the duration of the study
* In otherwise good health as determined by medical history, physical examination, results of screening tests and the clinical judgment of a medically qualified Clinical Investigator
* Negative for malaria on blood smear
* Judged, in the opinion of a medically qualified Clinical Investigator, to be able and likely to comply with all study requirements as set out in the protocol
* Willing to undergo screening for HIV, Hepatitis B and Hepatitis C
* Leishmania PCR positive on the screening skin biopsy
* For females only, willing to undergo urinary pregnancy tests on the day of screening, on the day of vaccination (prior to vaccination) and 7 and 42 days after vaccination.

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Has mucosal or conjunctival PKDL
* Has had treatment for PKDL within 21 days
* Receipt of a live attenuated vaccine within 60 days or other vaccine within 14 days of screening
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine or a history of severe or multiple allergies to drugs or pharmaceutical agents
* Any history of severe local or general reaction to vaccination as defined as
* Local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
* General: fever ≥ 39.5°C within 48 hours, anaphylaxis, bronchospasm, laryngeal oedema, collapse, convulsions or encephalopathy within 48 hours
* Females - pregnancy, less than 12 weeks postpartum, lactating or willingness/intention to become pregnant during the study and for 3 months following vaccination.
* Seropositive for hepatitis B surface antigen (HBsAg) or Hepatitis C (antibodies to HCV)
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months
* Tuberculosis, leprosy, or malnutrition (malnutrition in adults defined as a BMI <18.5, and in adolescents (12-17yrs) as a Z score cut-off value of <-2 SD).
* Any other significant disease, disorder or finding, which, in the opinion of a medically qualified Clinical Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study
* Unlikely to comply with the study protocol

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
To assess the number of participants with treatment-related adverse events as defined in the clinical trial protocol V1.0. | 24 months
  To assess the number of participants with treatment-related adverse events as defined in the clinical trial protocol V1.0.
To assess the therapeutic efficacy of CHAd63-KH, a new candidate, in patients with PKDL by clinical judgement of PKDL lesion reduction. | 24 months
  To assess the therapeutic efficacy of CHAd63-KH, a new candidate, in patients with PKDL by clinical judgement of PKDL lesion reduction.

SECONDARY OUTCOMES:
Immune responses by presence of interferon gamma producing T cells | 24 months
  To identify cellular immune responses generated by the candidate vaccine in patients with persistent PKDL using a gamma interferon ELISpot assay
Immune responses by presence of serum antibodies against Leishmania peptides | 24 months
  To identify humoral immune responses generated by the candidate vaccine in patients with persistent PKDL using a gamma interferon ELISpot assay
Clinical changes in PKDL disease | 24 months
  To observe any changes in the appearance of the cutaneous PKDL disease over a 120 day period following vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Tropical Medicine, Doka, Gedarif, Sudan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Younis BM, Wiggins R, Khalil EAG, Osman M, Santoro F, Sonnati C, Keding A, Novedrati M, Montesi G, Noureldein A, Elmukashfi ETA, Mustafa AE, Alamin M, Saeed M, Salman K, Suliman AJ, Musa AEA, Layton AM, Lacey CJN, Kaye PM, Musa AM. A randomized, double-blind phase 2b trial to evaluate efficacy of ChAd63-KH for treatment of post kala-azar dermal leishmaniasis. Mol Ther Methods Clin Dev. 2024 Jul 30;32(3):101310. doi: 10.1016/j.omtm.2024.101310. eCollection 2024 Sep 12. PMID 39253357
- [Derived] Lacey C, Musa A, Khalil ET, Younis B, Osman M, Wiggins R, Keding A, Kaye P. LEISH2b - A phase 2b study to assess the safety, efficacy, and immunogenicity of the Leishmania vaccine ChAd63-KH in post-kala azar dermal leishmaniasis. Wellcome Open Res. 2022 Aug 3;7:200. doi: 10.12688/wellcomeopenres.17951.1. eCollection 2022. PMID 37252616